CLINICAL TRIAL: NCT01818193
Title: Neurological Complications - Pulmonary Transplant
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/60
Record Dates: First submitted 2013-03-13; First posted 2013-03-26 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Cognitive Dysfunctions
Keywords: Pulmonary transplant
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A monocentric prospective open study to evaluate the frequency and nature of cognitive complications in the 3rd month post pulmonary transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years of age.
* Enregistered in lung transplant waiting list
* Have given their agreement to be enrolled in the study

Exclusion Criteria:

* Patients had a previous lung transplant
* patients with insufficient level of french language that may affect the comprehension and answering the psychometric test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enregistered in the waiting list for lung transplant
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rey auditory verbal learning test | 3 months
Rey complex figure test | 3 months
Boston naming test of 30 figures | 3 months
Visual construction skills | 3 months
Grooved Pegboard test | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital FOCH, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No